CLINICAL TRIAL: NCT06574178
Title: Use of Total-Body PET to Quantify Systemic and Cutaneous Inflammation in Psoriasis Patients Before and After Intervention With a Nutritionally Balanced Diet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1912111
Record Dates: First submitted 2024-08-15; First posted 2024-08-27 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Psoriasis
Keywords: western diet; Total-body PET
MeSH Terms: conditions — Psoriasis | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary Intervention (Experimental): Participants will receive breakfast, lunch, and dinner in the form of fully cooked, ready-to-heat standardized meals for 6 weeks that are prepared by a commercial kitchen.
  Interventions: Behavioral: Dietary Counseling

INTERVENTIONS:
Behavioral: Dietary Counseling — A Registered Dietitian or Nutritionist will provide nutrition education either in person, over the phone, or via Zoom. The behavioral program will use cognitive-behavioral techniques to foster adherence to diet prescriptions and to build a supportive environment for the participant.

SUMMARY:
Psoriasis is a chronic inflammatory disease that affects the skin and joints in 2-3 % of people in the United States. This inflammation of the skin, joints, and blood vessels in patients with psoriasis has been measured by older PET Scan technology but with limitations. With the new EXPLORER PET scanner technology, the investigators are testing to see if the EXPLORER is better than previous PET scanners and improve our ability to assess inflammation in patients.

Also, it is known that the typical Western Diet - high in saturated fats, added sugars, and low in fiber - contributes to obesity and inflammation worldwide. There is evidence in animals that these signs of inflammation are reversible within 4 weeks when changed to a more balanced diet. Thus, this study aims to assess whether there are detectable decreases in inflammation of the skin and body of psoriasis patients who usually eat a Western Diet on an EXPLORER PET scan following 6 weeks of a more balanced diet.

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory disease that affects the skin and joints of up to 2-3% of the US population and well known to be associated with multiple medical co-morbidities, including cardiac disease, type 2 diabetes, and obesity. Skin, joint, vascular and organ inflammation has been measured in patients with psoriasis using older PET imaging methodologies4,5 and correlated with disease6. The Hwang lab has shown that mice triggered with systemic exposure to IL-23, a known pathogenic cytokine in human psoriasis, will develop PET-detectable signs of inflammation in joints, and, that this PET signal is greatly diminished by an antagonist of CCR6, a chemokine receptor believed to play a key role in Th17 cell migration7.

Dietary patterns containing high amounts of saturated fat, added sugars, and low in dietary fiber - also known as Western diet (WD)- are thought to be a major contributor to the epidemic of obesity worldwide. The Hwang lab has recently also shown that mice fed a WD show histologic, clinical, and molecular signs of psoriasis within 4 weeks8 which are accompanied by striking changes in the gut microbiome9. In addition, the WD accentuates IL-23-mediated skin and joint inflammation in mice, which is partially reversible when the animals are then placed on a conventional balanced diet9. Data from studies in humans support that weight loss may be an effective adjunct to medical treatment to ameliorate signs and symptoms of psoriasis, prompting the National Psoriasis Foundation to strongly recommend caloric restriction to achieve weight loss in obese psoriatic patients10. However, the role of diet composition/quality in psoriasis-related outcomes remains currently poorly understood. To this end, the overarching goal of this pilot study is to determine whether or not a 6-week dietary intervention that follows the current nutrition guidelines for chronic disease prevention (healthy diet)11-13 can affect psoriasis-related outcomes in patients with psoriasis who generally consume a WD.

These published studies lead us to hypothesize that dietary intervention, even in as little as 6 weeks, will reduce PET-measurable skin and systemic signs of inflammation in patients with psoriasis who habitually consume a WD that is high in fat and sugar content.

The EXPLORER scanner is unique because it has: (i) an axial field of view of 194 cm that covers the entire adult human body in a single bed position; (ii) increased detection efficiency (by a factor of ~40) for whole-body PET imaging compared to standard scanners, thus enabling dose reduction and/or faster scanning; and (iii) a PET spatial resolution (~3 mm) that significantly exceeds that of most current whole-body PET/CT scanners. The investigators believe that this technology has potential to overcome limitations of current PET/CT technology and significantly positively impact patient assessment.

Given the speed, whole-body coverage, and spatial resolution of the Total-body PET EXPLORER scanner at UC Davis, the investigators propose to test this hypothesis by quantitatively assessing uptake of 18F-FDG in recruited patients before dietary intervention and then 6 weeks later after intervention with a nutritionally recommended diet. Normal, healthy controls who have had previous scans performed under the same protocol will be available for comparative purposes. If several of the planned enrollment of 5 patients show demonstrable decreases in systemic inflammation, the preliminary pilot data will be vital to support an application for NIH R-type grant to explore the use of total-body PET imaging to assess systemic inflammation in psoriatic patients as well as to justify the clinical need for dietary interventions in what are considered autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 year)
* Both sexes
* Must have a history of psoriasis of at least 3% body surface area affected by skin psoriasis (in a body area that the subject will allow the PI to perform several skin biopsies as noted below (optional)) and may carry a diagnosis of psoriatic arthritis as well
* Patients will have a BMI of >/=25 which is consistent with being overweight - Willing and able to fast for at least 6 hours before and for the duration of the scan visit
* No strenuous exercise for 24 hours prior to being scanned
* Recruited patients must habitually consume a WD-type diet that will be evaluated by using DHQ III food frequency questionnaire along with three-day food record14. Subsequently, the Healthy Eating Index will be calculated and participants with a poor dietary pattern (score below 58) will be eligible for the study15.

Exclusion Criteria:

* Those taking anti-diabetic oral or injected medications
* Those already ingesting a caloric- or component-restricted diet
* Vegan, vegetarian or food allergy or intolerance to the ingredients of the diet
* >5% change in body weight in the last 2 months
* Those taking systemic medications for the purpose of treating psoriasis or psoriatic arthritis for at least 3 months prior to first PET scan or during the duration of the trial
* Self-reported history of dysphoria or anxiety in closed spaces (claustrophobia)
* Uncontrolled diabetes or blood glucose level greater than 180 mg/dl at the time of radiotracer injection
* Body weight >240 kg due to limitations of the scanner bed
* Known inflammatory or other infectious disease that can confound assessment
* Pregnant or breast-feeding (urine pregnancy test will be administered prior to start of each PET/CT session for all participants who are able to get pregnant between 18 to 60 years old, unless documented hysterectomy or bilateral ovarian removal is available, because of risks from ionizing radiation)
* Inability to lie motionless on the scanner bed with the arms by the side for up to 60 minutes
* Currently participating in another conflicting research study. Concurrent or prior enrollment in a separate research study involving a PET scan performed within the last 12 months for research purposes only.
* Unwilling to sign informed consent
* Inability to understand the risks and benefits of the study
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Inflammation in PET/CT scan | in Week 0 and Week 6
  measuring inflammation in PET imaging by calculating the maximum standardized uptake values (SUVmax) in given areas of interest (e.g., joint, blood vessel)

SECONDARY OUTCOMES:
Microbiomes Diversity | in Week 0 and Week 6
  Measuring changes in stool and skin microbiome both through alpha diversity analysis measured in operational taxonomic units, and through beta diversity analysis using unweighted UniFrac Distance Principal Coordinates Analysis Plots (Shi et al.,2021)
Serum Inflammatory Markers | in Week 0 and Week 6
  measuring TNF, IL-17A, and CRP levels through ELISA methods in blood samples
Cell Surface Inflammatory Markers | in Week 0 and Week 6
  measuring cell surface integrin, L-selectin, CD11b, and CD66b levels by standard flow cytometric methods in blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel T Hwang, MD, PhD, Principal Investigator — UC Davis SOM Department of Dermatology
Locations (1):
- University of California, Davis - Dermatology Department, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang X, Badawi RD, Cherry SR, Qi J. Theoretical study of the benefit of long axial field-of-view PET on region of interest quantification. Phys Med Biol. 2018 Jun 27;63(13):135010. doi: 10.1088/1361-6560/aac815. PMID 29799814
- [Background] Badawi R, Liu W, Berg E, et al. Progress on the EXPLORER project: towards a total body PET scanner for human imaging. J Nucl Med. 2018;59(supplement 1):223-223. http://jnm.snmjournals.org/content/59/supplement_1/223.short#cited-by.
- [Background] Cherry SR, Badawi RD, Karp JS, Moses WW, Price P, Jones T. Total-body imaging: Transforming the role of positron emission tomography. Sci Transl Med. 2017 Mar 15;9(381):eaaf6169. doi: 10.1126/scitranslmed.aaf6169. PMID 28298419
- [Background] Mehta NN, Yu Y, Saboury B, Foroughi N, Krishnamoorthy P, Raper A, Baer A, Antigua J, Van Voorhees AS, Torigian DA, Alavi A, Gelfand JM. Systemic and vascular inflammation in patients with moderate to severe psoriasis as measured by [18F]-fluorodeoxyglucose positron emission tomography-computed tomography (FDG-PET/CT): a pilot study. Arch Dermatol. 2011 Sep;147(9):1031-9. doi: 10.1001/archdermatol.2011.119. Epub 2011 May 16. PMID 21576552
- [Background] Chaudhari AJ, Ferrero A, Godinez F, Yang K, Shelton DK, Hunter JC, Naguwa SM, Boone JM, Raychaudhuri SP, Badawi RD. High-resolution (18)F-FDG PET/CT for assessing disease activity in rheumatoid and psoriatic arthritis: findings of a prospective pilot study. Br J Radiol. 2016 Jul;89(1063):20160138. doi: 10.1259/bjr.20160138. Epub 2016 Apr 25. PMID 27109738
- [Background] Naik HB, Natarajan B, Stansky E, Ahlman MA, Teague H, Salahuddin T, Ng Q, Joshi AA, Krishnamoorthy P, Dave J, Rose SM, Doveikis J, Playford MP, Prussick RB, Ehrlich A, Kaplan MJ, Lockshin BN, Gelfand JM, Mehta NN. Severity of Psoriasis Associates With Aortic Vascular Inflammation Detected by FDG PET/CT and Neutrophil Activation in a Prospective Observational Study. Arterioscler Thromb Vasc Biol. 2015 Dec;35(12):2667-76. doi: 10.1161/ATVBAHA.115.306460. Epub 2015 Oct 8. PMID 26449753
- [Background] Shi Z, Garcia-Melchor E, Wu X, Getschman AE, Nguyen M, Rowland DJ, Wilson M, Sunzini F, Akbar M, Huynh M, Law T, Raychaudhuri SK, Raychaudhuri SP, Volkman BF, Millar NL, Hwang ST. Targeting the CCR6/CCL20 Axis in Entheseal and Cutaneous Inflammation. Arthritis Rheumatol. 2021 Dec;73(12):2271-2281. doi: 10.1002/art.41882. Epub 2021 Nov 1. PMID 34081845
- [Background] Shi Z, Wu X, Yu S, Huynh M, Jena PK, Nguyen M, Wan YY, Hwang ST. Short-Term Exposure to a Western Diet Induces Psoriasiform Dermatitis by Promoting Accumulation of IL-17A-Producing gammadelta T Cells. J Invest Dermatol. 2020 Sep;140(9):1815-1823. doi: 10.1016/j.jid.2020.01.020. Epub 2020 Feb 10. PMID 32057839
- [Background] Shi Z, Wu X, Santos Rocha C, Rolston M, Garcia-Melchor E, Huynh M, Nguyen M, Law T, Haas KN, Yamada D, Millar NL, Wan YY, Dandekar S, Hwang ST. Short-Term Western Diet Intake Promotes IL-23-Mediated Skin and Joint Inflammation Accompanied by Changes to the Gut Microbiota in Mice. J Invest Dermatol. 2021 Jul;141(7):1780-1791. doi: 10.1016/j.jid.2020.11.032. Epub 2021 Jan 22. PMID 33485880
- [Background] Ford AR, Siegel M, Bagel J, Cordoro KM, Garg A, Gottlieb A, Green LJ, Gudjonsson JE, Koo J, Lebwohl M, Liao W, Mandelin AM 2nd, Markenson JA, Mehta N, Merola JF, Prussick R, Ryan C, Schwartzman S, Siegel EL, Van Voorhees AS, Wu JJ, Armstrong AW. Dietary Recommendations for Adults With Psoriasis or Psoriatic Arthritis From the Medical Board of the National Psoriasis Foundation: A Systematic Review. JAMA Dermatol. 2018 Aug 1;154(8):934-950. doi: 10.1001/jamadermatol.2018.1412. PMID 29926091
- [Background] Krauss RM, Eckel RH, Howard B, Appel LJ, Daniels SR, Deckelbaum RJ, Erdman JW Jr, Kris-Etherton P, Goldberg IJ, Kotchen TA, Lichtenstein AH, Mitch WE, Mullis R, Robinson K, Wylie-Rosett J, St Jeor S, Suttie J, Tribble DL, Bazzarre TL. AHA Dietary Guidelines: revision 2000: A statement for healthcare professionals from the Nutrition Committee of the American Heart Association. Circulation. 2000 Oct 31;102(18):2284-99. doi: 10.1161/01.cir.102.18.2284. No abstract available. PMID 11056107
- [Background] American Diabetes Association. 4. Lifestyle Management: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018 Jan;41(Suppl 1):S38-S50. doi: 10.2337/dc18-S004. PMID 29222375
- [Background] Subar AF, Thompson FE, Kipnis V, Midthune D, Hurwitz P, McNutt S, McIntosh A, Rosenfeld S. Comparative validation of the Block, Willett, and National Cancer Institute food frequency questionnaires : the Eating at America's Table Study. Am J Epidemiol. 2001 Dec 15;154(12):1089-99. doi: 10.1093/aje/154.12.1089. PMID 11744511
- [Background] Kennedy ET, Ohls J, Carlson S, Fleming K. The Healthy Eating Index: design and applications. J Am Diet Assoc. 1995 Oct;95(10):1103-8. doi: 10.1016/S0002-8223(95)00300-2. PMID 7560680
- [Background] Webb VL, Wadden TA. Intensive Lifestyle Intervention for Obesity: Principles, Practices, and Results. Gastroenterology. 2017 May;152(7):1752-1764. doi: 10.1053/j.gastro.2017.01.045. Epub 2017 Feb 10. PMID 28192109
- [Background] Williamson DA. Fifty Years of Behavioral/Lifestyle Interventions for Overweight and Obesity: Where Have We Been and Where Are We Going? Obesity (Silver Spring). 2017 Nov;25(11):1867-1875. doi: 10.1002/oby.21914. Epub 2017 Sep 25. PMID 28944593